CLINICAL TRIAL: NCT05376358
Title: Technology and Emotion Study "TECH-E": Randomized Controlled Trial of MoodRing Compared to Usual Care: Mobile Monitoring of Adolescent Depression Phase II
Brief Title: Evaluation of MoodRing on Improving the Quality of Depression Management in Adolescents
Acronym: TECH-E
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prior to being able to recruit the full sample due to lack of funding and expiration of time on the award. The sample recruited completed the entire 6 month study.
Sponsor: Ana Radovic (Other)
Collaborators: NuRelm, Inc. (Industry); National Institute of Mental Health (NIMH) (NIH); University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Ana Radovic, Assistant Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY21050120; R44MH122067 (NIH)
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Depression in Adolescence
Keywords: Adolescent; Adolescent Medicine; Mental Health Services; eHealth; Mobile Applications; Symptom Management

STUDY DESIGN:
Intervention Model Description: This study will use a parallel study design, where participants are randomized into two intervention groups (Usual Care or MoodRing) and will receive interventions in parallel.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to the intervention condition at follow-up assessment time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Participants in this arm will receive no intervention and access treatment as usual per their mental health services provider. A mobile application (AWARE) which is not interactive and is only for purposes of data collection will be downloaded on the adolescents' smartphone.
  Interventions: Other: Usual Care
- MoodRing (Experimental): Adolescent participants in this arm will download two mobile applications - a data collection non-interactive app to collect passive sensing data (AWARE) and the MoodRing (MR) mobile application with which they can visualize their data about their mood, sleep, activity, enter their own mood score, and access psychoeducational resources including links to a research-based website, SOVA. Their parents will download a parent MoodRing application which provides them with parenting resources and articles and a weekly report of their adolescents' mood as predicted by passive sensing. Clinical providers will receive access to a web portal where they can view their adolescent patients' data who are enrolled in the study.
  Interventions: Device: MoodRing App

INTERVENTIONS:
Device: MoodRing App — Adolescents and parents in the MR arm will receive instructions to download the MR app and AWARE app, customize the app, utilize an app-based self-guided onboarding, and review questions with the research team. The MR app provides the adolescent and their parent a notification to view a weekly report predicting their mood score (i.e. depression severity level similar to the Patient health questionnaire-9). The MR app will provide a library of coping strategies for adolescents and opportunities to self-track their mood.
  Clinicians in the MR Arm will get access to a MR portal online. They will be able to view patients they are a provider for. The clinician will receive in-person and/or video-based training to use the portal.
  Arms: MoodRing
Other: Usual Care — Adolescents and parents in the usual care arm will receive instructions to download the AWARE app. This app will only track data and will not be interactive. Otherwise they will receive care as per routine by their healthcare provider team.
  Arms: Usual Care

SUMMARY:
The MoodRing intervention is a mobile application for adolescents, parents, and an accompanying web-based clinician portal which enables adolescents to monitor their mood through the use of passively collected smartphone data. This randomized controlled trial will evaluate whether MoodRing as compared to usual care improves the quality of depression management.

DETAILED DESCRIPTION:
This is a randomized controlled trial to evaluate the efficacy of MoodRing as compared to usual care for adolescents who have a prior diagnosis of depression. Adolescents with depressive symptoms, their parents, and their mental healthcare providers (if interested) will participate in a 6 month study. Adolescents age 12-18 and their parent will be consented for the study and be sent an online survey to obtain baseline measures. Those who complete the baseline measures will then be randomized to receive the MoodRing intervention or treatment as usual. Adolescents and parents will be asked to complete data collection at 3 months and 6 month time points post-randomization by online survey. Additionally, data will be collected for 3 and 6 month timepoints via the adolescent's electronic health record data. At 6 months, online surveys will be sent and an invitation to interview for patients' mental healthcare providers who consent to participate in the study.

Adolescent-parent dyads will be randomized at a 1:1 ratio (using randomized block sizes) to either 1) MoodRing or 2) usual care. 100 adolescent-parent dyads (200 total individuals) will be randomized to MoodRing and 100 adolescent-parent dyads (200 total individuals) will be randomized to usual care. We expect 50 clinicians will participate. In both arms, passively collected data will be obtained from adolescent smartphones as well as weekly mood surveys and monthly sleep surveys. In the 1) MoodRing arm adolescents will download the MoodRing-adolescent app, parents will download the MoodRing-parent app, and healthcare providers if interested will have access to a clinician dashboard. The randomization tables will be generated by the study statistician.

The investigators hypothesize that adolescents who receive MoodRing as compared to usual care will have:

H1: Improved self-management of depression as measured by change of baseline for the average score on the Partners in Health Scale

EH2: The investigators will also explore whether MoodRing as compared to usual care will result in improved quality of depression management as measured by frequency of symptom reassessment, medication adherence, and therapy adherence, less healthcare utilization, decreased depression symptoms, improved sleep quality, and increased application of self-management activities through increased self-efficacy, utilization of self-management skills and knowledge and social support.

H3: The investigators anticipate healthcare providers, adolescents, and parents will report satisfaction with use of MoodRing.

* After date September 2022, we decided to make a change to the protocol and primary outcome. Due to recruitment challenges from mental health clinicians due to their clinical workload, we made a change to recruit adolescents directly including using social media. This introduced more heterogeneity to access to mental health care as well as less access to electronic health records systems that were external to our site which made it less likely to be able to measure quality of depression management. For this reason, the goal to recruit healthcare providers was discontinued. And the primary outcome was changed to self-management, changing our hypothesis to:

We hypothesized that MoodRing will help adolescents better self-manage their depression.

Secondary outcome measures were changed from "change in symptoms" to just that symptom total at 3 months and 6 months for better clinical interpretability.

ELIGIBILITY:
Inclusion Criteria:

Adolescent:

* age 12 -18
* prior or present history of depression per self-report and/or clinician diagnosis
* scores between 5 or higher on PHQ-9 consistent with at least mild symptoms of depression
* read and understand English
* has an Android or iOS smartphone compatible with AWARE mobile application and access to a smartphone data plan
* currently in United States

Parent/Guardian:

* adolescent qualifies for study and assents to enroll
* understands English
* currently in United States
* has a smartphone device that can download the intervention application

Healthcare Provider:

- involved in providing mental health treatment (psychotherapy or antidepressant prescribing or making referrals) to adolescent participant - can be a primary care provider, therapist, subspecialist, psychiatrist

Exclusion Criteria:

Adolescent:

* currently actively suicidal (have suicidal thoughts and plan with an intent to act on it)
* plans to travel to countries belonging to the European Union (Austria, Belgium, Bulgaria, Croatia, Cyprus, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Hungary, Ireland, Italy, Latvia, Lithuania, Luxembourg, Malta, The Netherlands, Poland, Portugal, Romania, Slovakia, Slovenia, Spain, Sweden), the United Kingdom (England, Scotland, Wales, and Northern Ireland), Norway, Iceland, or Lichtenstein in the next 6 months for more than 2 weeks at a time

Parent:

- If their adolescent child is excluded

Healthcare Provider:

- None

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Shaaban, BSEE, MBA, Principal Investigator — NuRelm, Inc.; Ana Radovic, MD, MSc, Principal Investigator — University of Pittsburgh; Afsaneh Doryab, Ph.D. CS, Principal Investigator — University of Virginia
Locations (1):
- Center for Adolescent and Young Adult Health, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Trial outcome data can be accessed by contacting the study principal investigator. Otherwise there is currently no formal plan for data sharing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment sources: 81.4% from social media advertisement (591/726), 9.5% completing an electronic interest form in clinic at UPMC Children's Hospital of Pittsburgh Center for Adolescent and Young Adult Health (69/726), and from 9% completing the University of Pittsburgh online interest form (Pitt+Me) (66/726). Out of these, 12.5% (91/726) were able to be reached to complete screening. Prior to the study a plan was made to enroll healthcare providers. One provider was approached did not enroll.
Pre-assignment Details: Both the adolescent and the parent were required to complete the baseline survey to enter the study. Out of 73 adolescent and parent dyads consented for the study, 68 (93.1%) of adolescents completed the baseline survey while, despite multiple contacts, only 63 (86.3%) of parents completed the baseline. Therefore 63 adolescent parent dyads were able to start the study and were randomized.
Groups:
- MoodRing: Adolescent participants in this arm will download two mobile applications - a data collection non-interactive app to collect passive sensing data (AWARE) and the MoodRing (MR) mobile application with which they can visualize their data about their mood, sleep, activity, enter their own mood score, and access psychoeducational resources including links to a research-based website, SOVA. Their parents will download a parent MoodRing application which provides them with parenting resources and articles and a weekly report of their adolescents' mood as predicted by passive sensing. Clinical providers will receive access to a web portal where they can view their adolescent patients' data who are enrolled in the study.
  MoodRing App: Adolescents and parents in the MR arm will receive instructions to download the MR app and AWARE app, customize the app, utilize an app-based self-guided onboarding, and review questions with the research team. The MR app provides the adolescent and their parent a notification to view a weekly report predicting their mood score (i.e. depression severity level similar to the Patient health questionnaire-9). The MR app will provide a library of coping strategies for adolescents and opportunities to self-track their mood.
  Clinicians in the MR Arm will get access to a MR portal online. They will be able to view patients they are a provider for. The clinician will receive in-person and/or video-based training to use the portal.
Period: 3 Month Timepoint Data Collection
Arm/Group | Usual Care | MoodRing
Started | 31 (31 Adolescents and 31 Parents) | 32 (32 adolescents and 32 parents)
Completed | 12 (12 dyads completed 3 month data collection) | 9 (9 dyads completed 3 month data collection)
Not Completed | 19 | 23
Not completed — Dyads who did not complete 3 month due to parent not completing (ONLY ADOLESCENT COMPLETED) | 13 | 15
Not completed — Dyads who did not complete 3 month due to adolescent not completing (ONLY PARENT COMPLETED) | 3 | 3
Not completed — Lost to Follow-up | 3 | 5
Period: 6 Month Timepoint Data Collection
Arm/Group | Usual Care | MoodRing
Started (each dyad was able to complete 6 month timepoint regardless of whether or not they completed the 3 month timepoint) | 31 | 32
Completed | 8 (8 dyads completed the 6 month timepoint) | 8 (8 dyads completed 6 month timepoint)
Not Completed | 23 | 24
Not completed — Dyads who did not complete 6 month due to parent not completing (ONLY ADOLESCENT COMPLETED) | 14 | 13
Not completed — Dyads who did not complete 6 month due to parent not completing (ONLY ADOLESCENT COMPLETED) | 1 | 5
Not completed — Lost to Follow-up | 8 | 6

BASELINE CHARACTERISTICS:
Population: For age: Adolescents and Parents are reported separately because providing a total average age across adolescents and parents is not indicated.
Groups:
- MoodRing - Adolescents: Adolescent participants in this arm will download two mobile applications - a data collection non-interactive app to collect passive sensing data (AWARE) and the MoodRing (MR) mobile application with which they can visualize their data about their mood, sleep, activity, enter their own mood score, and access psychoeducational resources including links to a research-based website, SOVA.
  MoodRing App: Adolescents in the MR arm will receive instructions to download the MR app and AWARE app, customize the app, utilize an app-based self-guided onboarding, and review questions with the research team. The MR app provides the adolescent a notification to view a weekly report predicting their mood score (i.e. depression severity level similar to the Patient health questionnaire-9). The MR app will provide a library of coping strategies for adolescents and opportunities to self-track their mood.
- MoodRing - Parents: Parents will download a parent MoodRing application which provides them with parenting resources and articles and a weekly report of their adolescents' mood as predicted by passive sensing. The MR app provides the parent a notification to view a weekly report predicting their mood score (i.e. depression severity level similar to the Patient health questionnaire-9).
- Usual Care - Adolescents: Participants in this arm will receive no intervention and access treatment as usual per their mental health services provider. A mobile application (AWARE) which is not interactive and is only for purposes of data collection will be downloaded on the adolescents' smartphone.
  Usual Care: Adolescents in the usual care arm will receive instructions to download the AWARE app. This app will only track data and will not be interactive. Otherwise they will receive care as per routine by their healthcare provider team.
- Usual Care - Parents: Parents will not receive an intervention but only complete data collection.
- Total: Total of all reporting groups
Arm/Group | MoodRing - Adolescents | MoodRing - Parents | Usual Care - Adolescents | Usual Care - Parents | Total
Number analyzed (Participants) | 32 | 32 | 31 | 31 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: When calculating average adolescent age, 0 parent participants were analyzed. When calculating average parent age, 0 adolescent participants were analyzed.
  years
    Adolescents: number analyzed (Participants) | 32 | 0 | 31 | 0 | 63
    Adolescents | 16.25 (1.41) |  | 15.65 (1.45) |  | 15.95 (1.43)
    Parents: number analyzed (Participants) | 0 | 32 | 0 | 31 | 63
    Parents |  | 45.12 (6.8) |  | 47.16 (7.08) | 46.12 (6.94)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Boy/Man | 8 | 2 | 10 | 0 | 20
  Girl/Woman | 18 | 30 | 19 | 31 | 98
  Not applicable | 6 | 0 | 2 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 4 | 2 | 8
  Not Hispanic or Latino | 30 | 32 | 27 | 29 | 118
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 1 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 3 | 2 | 3 | 11
  White | 23 | 26 | 23 | 26 | 98
  More than one race | 3 | 0 | 4 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Self-Management [Mean (Standard Deviation); unit: units on a scale] — Partners in Health Scale The revised Partners in Health Scale (Smith 2016) assesses self-management with respect to a chronic condition, with regard to active involvement of a patient in managing their condition. Total scores range from 0 to 96 with higher scores indicating worse self-management. Population: parents were not asked this measure
  units on a scale
    number analyzed (Participants) | 32 | 0 | 31 | 0 | 63
    (all) | 60.72 (18.14) |  | 59.74 (13.51) |  | 60.24 (15.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Self-management at 3 Months
Description: Adolescents will be asked the Partners in Health Scale The revised Partners in Health Scale (Smith 2016) assesses self-management with respect to a chronic condition, with regard to active involvement of a patient in managing their condition. Total scores range from 0 to 96 with higher scores indicating worse self-management.
  A larger negative change in self-management score means an improvement in self-management.
Time Frame: From baseline to 3 months
Population: The pre-specified statistical analysis was not scientifically appropriate due to insufficient enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
score on a scale | 12 (14.3) | -1.84 (16.04)

2. Secondary Outcome: Quality of Depression Management: Depression Symptom Reassessment
Description: Attendance at a healthcare provider visit for depression symptom reassessment within 3 months (yes/no) measured by adolescent or parent self-report (yes if any are yes, no if all are no). The metric reported will be percentage of individuals per study arm with a 'yes' result.
Time Frame: 3 months
Population: Number participants include Adolescents who did not respond to the question on their baseline survey but their Parents did - total number of responses measured by adolescent or parent self-report even if one was missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 29 | 28
Participants | 20 | 24

3. Secondary Outcome: Quality of Depression Management: Medication Adherence
Description: Out of adolescents who are taking an antidepressant, receipt of at least 60 consecutive days (yes/no) measured by adolescent self-report. The metric reported will be percentage of individuals per study arm with a 'yes' result.
Time Frame: 3 months
Population: Number analyzed are adolescents who either themselves or their parent indicate taking/being prescribed an antidepressant.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 16 | 16
Participants | 16 | 12

4. Secondary Outcome: Quality of Depression Management: Therapy Adherence
Description: Out of adolescents who report being referred for psychotherapy, receipt of at least 3 sessions within 3 months (yes/no) measured by adolescent and parent self-report (yes if any are yes, no if all are no). The metric reported will be percentage of individuals per study arm with a 'yes' result.
Time Frame: 3 months
Population: Number analyzed were adolescents who either themselves or had their parent indicate that they were referred for psychotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 18 | 16
Participants | 15 | 14

5. Secondary Outcome: Healthcare Utilization for Acute Care or Primary Care (for Non Mental-health Reason)
Description: Average Number of visits for (greater number as reported by adolescent self-report and parent self-report):
  1. urgent care;
  2. emergency room;
  3. inpatient hospitalization;
  4. acute primary care provider visit for non-mental health related concern;
  5. medical subspecialist visit
  6. surgical subspecialist visit
Time Frame: 3 month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: average number of visits
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 29 | 27
average number of visits
  Urgent Care Visits | 0.21 (0.53) | 0.20 (0.48)
  Emergency Room | 0.10 (0.31) | 0.22 (0.54)
  Inpatient Hospitalization | 0.10 (0.39) | 0 (0)
  Acute PCP visit non mental health | 0.52 (0.79) | 0.44 (0.95)
  Medical Subspecialist Visit | 0.62 (0.94) | 0.37 (0.71)
  Surgical Subspecialist Visit | 0.15 (0.46) | 0.15 (0.53)

6. Secondary Outcome: Depression Severity at 3 Months
Description: Adolescents will be asked the PHQ-9 Patient Health Questionnaire-9 measures depression severity with a score ranging from 0 to 27, a higher score indicating greater severity.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
score on a scale | 11.19 (3.56) | 11.17 (5.14)

7. Secondary Outcome: Sleep-Related Impairment at 3 Months
Description: Adolescents will respond to the PROMIS Pediatric Sleep-Related Impairment scale. This scale has four questions with response options of never, almost never, sometimes, almost always, and always, ranges from 4 to 19 with higher scores indicating higher levels of sleep-related impairment.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
score on a scale | 13.12 (3.85) | 13.17 (3.81)

8. Secondary Outcome: Sleep Disturbance at 3 Months
Description: Adolescents will respond to the PROMIS Pediatric Sleep Disturbance scale. This scale has four questions, the second (sleeping through the night) being reverse-scored, with response options of never, almost never, sometimes, almost always, and always, ranges from 4 to 20 with higher scores indicating higher levels of sleep disturbance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
score on a scale | 13.48 (2.74) | 13.67 (3.67)

9. Secondary Outcome: Self-Efficacy at 3 Months
Description: Adolescents will be asked the Mental Health Self-efficacy Scale (MHSES) The Mental Health Self-efficacy Scale (Clarke, 2014) measures one's belief in one's capability to perform mental health self-care behaviors. The score ranges from 6 to 60, with higher scores indicating higher confidence in mental health selfcare.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
score on a scale | 33.62 (9.43) | 35.72 (9.77)

10. Secondary Outcome: Self-management Behavior at 3 Months
Description: Adolescents will be asked based on Question 12 of Partners in Health Scale about self-management behavior. This question asks the average amount of time (options including Daily, More than once a week, Once a week, Once a month, Once a semester, Once a year, Less than once a year, Never) spent in potentially useful self-management activities. Each time category will be described by a percentage. Each of the following are asked individually: (1) created to-do lists to help me focus; (2) found strategies to create pleasurable distractions; (3) engaged in some physical activity (cycling, walking, etc.); (4) set realistic short-term goals; (5) made sure I had a good day/night routine with got enough sleep; (6) ensured enough rest to avoid getting exhausted; (7) left the house regularly; (8) ate healthy
  A higher score indicates a better outcome.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
Participants
  Created to-do lists to help me focus: Daily | 4 | 5
  Created to-do lists to help me focus: More than Once a Week | 3 | 3
  Created to-do lists to help me focus: Once a Week | 3 | 5
  Created to-do lists to help me focus: Once a month | 7 | 0
  Created to-do lists to help me focus: Once a semester (3-4 months) | 4 | 3
  Created to-do lists to help me focus: Once a year | 1 | 3
  Created to-do lists to help me focus: Less than once a year | 4 | 0
  Created to-do lists to help me focus: Never | 0 | 6
  Found strategies to create pleasurable distractions: Daily | 2 | 5
  Found strategies to create pleasurable distractions: More than Once a Week | 7 | 6
  Found strategies to create pleasurable distractions: Once a Week | 9 | 3
  Found strategies to create pleasurable distractions: Once a month | 3 | 7
  Found strategies to create pleasurable distractions: Once a semester (3-4 months) | 3 | 2
  Found strategies to create pleasurable distractions: Once a year | 1 | 1
  Found strategies to create pleasurable distractions: Less than once a year | 1 | 1
  Found strategies to create pleasurable distractions: Never | 0 | 0
  Engaged in some moderate physical activity (cycling, walking, etc.): Daily | 2 | 11
  Engaged in some moderate physical activity (cycling, walking, etc.): More than Once a Week | 8 | 1
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a Week | 9 | 10
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a month | 4 | 2
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a semester (3-4 months) | 2 | 1
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a year | 0 | 0
  Engaged in some moderate physical activity (cycling, walking, etc.): Less than once a year | 1 | 0
  Engaged in some moderate physical activity (cycling, walking, etc.): Never | 0 | 0
  Set realistic short-term goals: Daily | 2 | 4
  Set realistic short-term goals: More than Once a Week | 5 | 3
  Set realistic short-term goals: Once a Week | 1 | 7
  Set realistic short-term goals: Once a month | 7 | 2
  Set realistic short-term goals: Once a semester (3-4 months) | 9 | 2
  Set realistic short-term goals: Once a year | 2 | 2
  Set realistic short-term goals: Less than once a year | 0 | 2
  Set realistic short-term goals: Never | 0 | 3
  Made sure I had a good day/night routine and got enough sleep: Daily | 1 | 4
  Made sure I had a good day/night routine and got enough sleep: More than Once a Week | 10 | 8
  Made sure I had a good day/night routine and got enough sleep: Once a Week | 5 | 6
  Made sure I had a good day/night routine and got enough sleep: Once a month | 3 | 2
  Made sure I had a good day/night routine and got enough sleep: Once a semester (3-4 months) | 4 | 3
  Made sure I had a good day/night routine and got enough sleep: Once a year | 2 | 0
  Made sure I had a good day/night routine and got enough sleep: Less than once a year | 0 | 2
  Made sure I had a good day/night routine and got enough sleep: Never | 1 | 0
  Ensured enough rest to avoid getting exhausted: Daily | 2 | 2
  Ensured enough rest to avoid getting exhausted: More than Once a Week | 7 | 8
  Ensured enough rest to avoid getting exhausted: Once a Week | 9 | 6
  Ensured enough rest to avoid getting exhausted: Once a month | 1 | 5
  Ensured enough rest to avoid getting exhausted: Once a semester (3-4 months) | 4 | 1
  Ensured enough rest to avoid getting exhausted: Once a year | 2 | 1
  Ensured enough rest to avoid getting exhausted: Less than once a year | 0 | 1
  Ensured enough rest to avoid getting exhausted: Never | 1 | 1
  Left the house regulary: Daily | 5 | 9
  Left the house regulary: More than Once a Week | 12 | 10
  Left the house regulary: Once a Week | 5 | 2
  Left the house regulary: Once a month | 3 | 1
  Left the house regulary: Once a semester (3-4 months) | 0 | 0
  Left the house regulary: Once a year | 1 | 1
  Left the house regulary: Less than once a year | 0 | 1
  Left the house regulary: Never | 0 | 1
  Ate healthy: Daily | 4 | 3
  Ate healthy: More than Once a Week | 14 | 12
  Ate healthy: Once a Week | 5 | 4
  Ate healthy: Once a month | 1 | 2
  Ate healthy: Once a semester (3-4 months) | 0 | 2
  Ate healthy: Once a year | 1 | 0
  Ate healthy: Less than once a year | 0 | 1
  Ate healthy: Never | 1 | 1

11. Secondary Outcome: Social Support at 3 Months
Description: Adolescents will be asked the Medical Outcomes Study Social Support Survey The Medical Outcome Study Social Support Scale (Sherbourne, 1991) measures types of social support. Each item ranges from 1 to 5 and the total score is averaged and ranges from 1 to 5, with higher levels associated with greater support.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 25
score on a scale | 3.66 (0.84) | 4.08 (0.72)

12. Secondary Outcome: Change in Self-management at 6 Months
Description: as for outcome 1
Time Frame: From baseline to 6 months
Population: Only participants completing this measure were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 20 | 20
score on a scale | -1.55 (13.3) | -4.6 (16.2)

13. Secondary Outcome: Quality of Depression Management: Depression Symptom Reassessment
Description: Attendance at a healthcare provider visit for depression symptom reassessment within the past 3 months (yes/no) measured by adolescent, parent self-report and electronic health record review (yes if any are yes, no if all are no). The metric reported will be percentage of individuals per study arm with a 'yes' result.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 22 | 25
Participants | 14 | 16

14. Secondary Outcome: Quality of Depression Management: Medication Adherence
Description: Out of adolescents who are taking an antidepressant, receipt of at least 60 consecutive days (yes/no) within the past 3 months, measured by adolescent, parent self-report and electronic health record review (yes if any are yes, no if all are no). The metric reported will be percentage of individuals per study arm with a 'yes' result.
Time Frame: 6 months
Population: Number analyzed were adolescents who either themselves or had their parent indicate that they are taking/prescribed an antidepressant.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 12 | 12
Participants | 11 | 11

15. Secondary Outcome: Quality of Depression Management: Therapy Adherence
Description: Out of adolescents who are referred for psychotherapy, receipt of at least 3 sessions within the past 3 months (yes/no) measured by adolescent, parent self-report and electronic health record review (yes if any are yes, no if all are no). The metric reported will be percentage of individuals per study arm with a 'yes' result.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 12 | 18
Participants | 11 | 17

16. Secondary Outcome: Healthcare Utilization for Acute Care or Primary Care (for Non Mental-health Reason)
Description: Number of visits for (combined total between adolescent self-report, parent self-report, and electronic health-record review):
  1. urgent care;
  2. emergency room;
  3. inpatient hospitalization;
  4. acute primary care provider visit for non-mental health related concern;
  5. medical or surgical subspecialist visit
Time Frame: 6 month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: patient visits
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 23 | 26
patient visits
  Urgent Care Visits | 0.22 (0.58) | 0.27 (0.64)
  Emergency Room | 0 (0) | 0.15 (0.43)
  Inpatient Hospitalization | 0 (0) | 0.04 (0.20)
  Acute PCP visit non mental health | 0.30 (0.52) | 0.27 (0.56)
  Medical Subspecialist Visit | 0.61 (1.19) | 0.94 (1.58)
  Surgical Subspecialist Visit | 0.13 (0.43) | 0.15 (0.54)

17. Secondary Outcome: Depression Severity at 6 Months
Description: as for outcome 6
Time Frame: 6 months
Population: Adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 26 | 24
score on a scale | 11.1 (4.88) | 8.45 (3.75)

18. Secondary Outcome: Self-management Behavior at 6 Months
Description: Adolescents will be asked based on Question 12 of Partners in Health Scale about self-management behavior. This question asks the average amount of time (options including Daily, More than once a week, Once a week, Once a month, Once a semester, Once a year, Less than once a year, Never) spent in potentially useful self-management activities. Each of the following are asked individually: (1) created to-do lists to help me focus; (2) found strategies to create pleasurable distractions; (3) engaged in some physical activity (cycling, walking, etc.); (4) set realistic short-term goals; (5) made sure I had a good day/night routine with got enough sleep; (6) ensured enough rest to avoid getting exhausted; (7) left the house regularly; (8) ate healthy
Time Frame: 6 months
Population: Adolescents
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 20 | 20
Participants
  to help me focus: Daily | 3 | 5
  to help me focus: More than Once a Week | 2 | 3
  to help me focus: Once a Week | 6 | 1
  to help me focus: Once a month | 3 | 3
  to help me focus: Once a semester (3-4 months) | 3 | 2
  to help me focus: Once a year | 0 | 3
  to help me focus: Less than once a year | 2 | 2
  to help me focus: Never | 1 | 1
  Found strategies to create pleasurable distractions: Daily | 3 | 7
  Found strategies to create pleasurable distractions: More than Once a Week | 4 | 5
  Found strategies to create pleasurable distractions: Once a Week | 7 | 3
  Found strategies to create pleasurable distractions: Once a month | 3 | 4
  Found strategies to create pleasurable distractions: Once a semester (3-4 months) | 2 | 0
  Found strategies to create pleasurable distractions: Once a year | 0 | 1
  Found strategies to create pleasurable distractions: Less than once a year | 1 | 0
  Found strategies to create pleasurable distractions: Never | 0 | 0
  Engaged in some moderate physical activity (cycling, walking, etc.): Daily | 6 | 6
  Engaged in some moderate physical activity (cycling, walking, etc.): More than Once a Week | 5 | 4
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a Week | 3 | 7
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a month | 5 | 1
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a semester (3-4 months) | 1 | 1
  Engaged in some moderate physical activity (cycling, walking, etc.): Once a year | 0 | 1
  Engaged in some moderate physical activity (cycling, walking, etc.): Less than once a year | 0 | 0
  Engaged in some moderate physical activity (cycling, walking, etc.): Never | 0 | 0
  Set realistic short-term goals: Daily | 2 | 5
  Set realistic short-term goals: More than Once a Week | 4 | 4
  Set realistic short-term goals: Once a Week | 2 | 6
  Set realistic short-term goals: Once a month | 4 | 2
  Set realistic short-term goals: Once a semester (3-4 months) | 5 | 2
  Set realistic short-term goals: Once a year | 2 | 1
  Set realistic short-term goals: Less than once a year | 0 | 0
  Set realistic short-term goals: Never | 1 | 0
  Made sure I had a good day/night routine and got enough sleep: Daily | 2 | 3
  Made sure I had a good day/night routine and got enough sleep: More than Once a Week | 3 | 7
  Made sure I had a good day/night routine and got enough sleep: Once a Week | 5 | 6
  Made sure I had a good day/night routine and got enough sleep: Once a month | 6 | 2
  Made sure I had a good day/night routine and got enough sleep: Once a semester (3-4 months) | 3 | 1
  Made sure I had a good day/night routine and got enough sleep: Once a year | 0 | 0
  Made sure I had a good day/night routine and got enough sleep: Less than once a year | 0 | 0
  Made sure I had a good day/night routine and got enough sleep: Never | 1 | 1
  Ensured enough rest to avoid getting exhausted: Daily | 3 | 1
  Ensured enough rest to avoid getting exhausted: More than Once a Week | 5 | 7
  Ensured enough rest to avoid getting exhausted: Once a Week | 2 | 8
  Ensured enough rest to avoid getting exhausted: Once a month | 7 | 2
  Ensured enough rest to avoid getting exhausted: Once a semester (3-4 months) | 2 | 0
  Ensured enough rest to avoid getting exhausted: Once a year | 0 | 1
  Ensured enough rest to avoid getting exhausted: Less than once a year | 1 | 0
  Ensured enough rest to avoid getting exhausted: Never | 0 | 1
  Left the house regularly: Daily | 4 | 10
  Left the house regularly: More than Once a Week | 11 | 6
  Left the house regularly: Once a Week | 5 | 2
  Left the house regularly: Once a month | 0 | 1
  Left the house regularly: Once a semester (3-4 months) | 0 | 1
  Left the house regularly: Once a year | 0 | 0
  Left the house regularly: Less than once a year | 0 | 0
  Left the house regularly: Never | 0 | 0
  Ate healthy: Daily | 5 | 3
  Ate healthy: More than Once a Week | 6 | 9
  Ate healthy: Once a Week | 6 | 4
  Ate healthy: Once a month | 2 | 1
  Ate healthy: Once a semester (3-4 months) | 0 | 2
  Ate healthy: Once a year | 1 | 1
  Ate healthy: Less than once a year | 0 | 0
  Ate healthy: Never | 0 | 0

19. Secondary Outcome: Self-Efficacy at 6 Months
Description: as for outcome 9
Time Frame: 6 months
Population: Adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 20 | 20
score on a scale | 37.5 (9.32) | 39.95 (10.56)

20. Secondary Outcome: Social Support at 6 Months
Description: as for outcome 11
Time Frame: 6 months
Population: Adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 20 | 20
score on a scale | 4.03 (0.76) | 4.04 (0.83)

21. Secondary Outcome: Sleep-Related Impairment at 6 Months
Description: as for outcome 7
Time Frame: 6 months
Population: Adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 20 | 20
score on a scale | 12.9 (4.79) | 13.05 (3.02)

22. Secondary Outcome: Sleep Disturbance at 6 Months
Description: as for outcome 8
Time Frame: 6 months
Population: Adolescent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | MoodRing
Number analyzed (Participants) | 20 | 20
score on a scale | 13.1 (2.63) | 13.65 (2.28)

23. Other Pre Specified Outcome: Sleep Habits at 3 Months
Description: Adolescents will respond to the School Based Sleep Habits Survey-Child Form which asks 43 questions about weekday and weeknight sleep patterns, sleep awakenings, and sleep time preferences.
Time Frame: 3 months
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Perceived Need for Service Use at 3 Months
Description: The General-practice Users Perceived-need Inventory (GUPI) The General-Practice Users Perceived-Need Inventory (McNab, 2004) will be used to measure perceived need for treatment. There is no scoring. Adolescents will be asked this and parents about their perception of their adolescent's need for mental health services. The response will be evaluated by the total number of individuals who agree that they would like to or are already getting help with a) medication and b) counseling as comapred to those who respond they do not need this kind of help.
Time Frame: 3 months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Perceived Severity at 3 Months
Description: Rating scale of General Mental Health A rating scale of General Mental Health (Cadigan, 2018) will be used with two questions each ranging from 1 to 5 with regard to a self-rating of general mental health. Adolescents will be asked this and parents about their perception of their adolescent's mental health.
Time Frame: 3 months
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Anxiety Severity at 3 Months
Description: Adolescents will be asked the GAD-7 Generalized Anxiety Disorders 7-item Questionnaire measures extent of anxiety symptoms. The total score ranges from 0 to 21 with a higher score indicating greater severity.
Time Frame: 3 months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Parent-Teen Communication Quality at 3 Months
Description: M-PACS (The Parent-Adolescent Communication Scale (Olson, 1985) modified for mental health) asks 20 questions with regards to communication between parents and adolescents, with responses 1-5 from strongly disagree to strongly agree. Some items are reverse scored with a higher scale score indicating better communication. Both adolescents and parents will be asked these questions.
Time Frame: 3 months
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Parent-Teen Relationship Quality at 3 Months
Description: The CPCS (Child Parent Connectedness Scale) asks 5 questions from a scale of 1-5 from strongly disagree to strongly agree with regards to connectedness and relationship satisfaction with each other. A higher score indicates higher child-parent connectedness. Both adolescents and parents will be asked these questions.
Time Frame: 3 months
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Suicidal Thoughts
Description: Adolescents who respond with anything besides "none" to the 9th question of the PHQ-9 will be asked to complete the brief CSSR-S scale. This scale asks two questions, have you (the participant) wished you (the participant) were dead or wished you (the participant) could go to sleep and not wake up? (yes/no) and have you (the participant) actually had any thoughts of killing yourself? (yes/no). Positive answers indicate suicidal thinking. These will be asked on an online survey. Those adolescents responding positively will complete a full CSSR-S interview.
Time Frame: 3 months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Sleep Habits at 6 Months
Description: as for outcome 23
Time Frame: 6 months
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Perceived Severity at 6 Months
Description: as for outcome 25
Time Frame: 6 months
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Perceived Need for Service Use at 6 Months
Description: as for outcome 24
Time Frame: 6 months
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Acceptability of MoodRing: Heathcare Provider Acceptability
Description: System Usability Questionnaire (Bangor, 2008) asks 11 questions about the usability of a technological intervention. SUS scores range from 0-100. Higher scores indicate better usability.
Time Frame: at 6 months
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Acceptability of MoodRing as a Clinical Tool: Heathcare Provider Acceptability
Description: Acceptability of Intervention Measure (AIM) (Weiner, 2017) asks 4 questions on a 1-5 Likert scale with completely disagree to completely agree with regards to acceptability of an intervention and 3 questions were added including with regards to efficiency, help taking care of patients, patient benefit from the intervention. Higher scores indicate higher acceptability. Also an open-ended question will be asked about feedback using MoodRing.
Time Frame: at 6 months
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Acceptability of MoodRing: Adolescent/Parent Acceptability
Description: System Usability Questionnaire (Bangor, 2008) asks 11 questions about the usability of a technological intervention. SUS scores 0-100. Higher scores indicate better usability. Adolescents and Parents - only those randomized to the MoodRing arm - will be asked these questions.
Time Frame: at 6 months
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Acceptability of MoodRing as a Self-management Tool: Adolescent/Parent Acceptability
Description: Acceptability of Intervention Measure (AIM) (Weiner, 2017) asks 4 questions on a 1-5 Likert scale with completely disagree to completely agree with regards to acceptability of an intervention. Additional questions will be asked about perceived benefit, taking care of mental health, and confidence in mental health management. Higher scores indicate higher acceptability. Also an open-ended question will be asked about feedback using MoodRing. Adolescents and Parents - only those randomized to the MoodRing arm - will be asked these questions.
Time Frame: at 6 months
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Anxiety Severity at 6 Months
Description: as for outcome 26
Time Frame: 6 months
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Parent-Teen Communication Quality at 6 Months
Description: as for outcome 27
Time Frame: 6 months
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Parent-Teen Relationship Quality at 6 Months
Description: as for outcome 28
Time Frame: 6 months
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Suicidal Thoughts
Description: as for outcome 29
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: This study was minimal risk. We did not actively assess for adverse events but had a plan to address if they were to spontaneously occur or be brought up by study participants. We monitored suicidality at 3 and 6 month time points and this was not assessed as an adverse event due to it being a part of the mental illness for some of the adolescents with depression in this trial.
Arm/Group | Usual Care | MoodRing
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 0/62 | 0/64

LIMITATIONS AND CAVEATS:
The pre-specified statistical analysis plan was not performed as it was not scientifically appropriate due to insufficient enrollment. Due to the complexity of intervention development and the COVID-19 pandemic we were not able to complete our enrollment goals prior to funding ceasing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT05376358/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT05376358/ICF_000.pdf